CLINICAL TRIAL: NCT02539498
Title: Characterization of Bone Architectural Parameters Assessed by High-Resolution Peripheral Quantitative Computed Tomography in Post-menopausal Women Affected With Primary Hyperparathyroidism
Brief Title: Bone Architectural Parameters in Postmenopausal Women Affected With Primary Hyperparathyroidism
Acronym: MicrOs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P091113
Record Dates: First submitted 2015-04-27; First posted 2015-09-03 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Primary Hyperparathyroidism; Bone Disease
Keywords: Primary Hyperparathyroidism; Parathyroid Hormone; High-Resolution peripheral Quantitative Computed Tomography; Bone densitometry; Bone microarchitecture
MeSH Terms: conditions — Hyperparathyroidism, Primary; Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Control post menopausal women without PHPT
  Interventions: Device: HR-pQCT
- Experimental (Experimental): Post menopausal women with PHPT followed for one year
  Interventions: Device: HR-pQCT

INTERVENTIONS:
Device: HR-pQCT — HR-pQCT to evaluate cortical and trabecular bone

SUMMARY:
Bone lesions are frequent in primary hyperparathyroidism (PHPT). Conventional measurement by Dual-Energy X-ray Absorptiometry does not provide enough information about the bone impact of excessive parathyroid hormone (PTH) secretion. High-Resolution peripheral Quantitative Computed Tomography (HR-pQCT) assesses separately cortical and trabecular bone sites as well as geometric characteristics of peripheral skeleton. In postmenopausal women, HR-pQCT has shown that decreased microarchitectural parameters are associated with reduced bone strength independently of BMD. The purpose of this study is to characterize the impact of PHPT in cortical and trabecular bone measured by HR-pQCT in postmenopausal women with PHPT followed for one year, in comparison with control postmenopausal women.

DETAILED DESCRIPTION:
Principal objective : To characterize the impact of PHPT in cortical and trabecular bone measured by HR-pQCT in postmenopausal women with PHPT followed for one year, in comparison with control postmenopausal women.

Secondary Objectives : 1) To compare the changes of bone micro-architecture in PHPT women with and without surgery to those of controls 2) To determine if the changes of micro-architecture are related to the severity of PTH secretion and to their changes after surgery 3) to evaluate the association of clinical and biological factors with quantitative bone micro-architectural indices and their changes.

Principal evaluation criteria : Cortical thickness

Secondary evaluation criteria : Quantitative parameters measured with HR-pQCT: trabecular microarchitecture (trabecular bone volume, number, separation, thickness and heterogeneity of trabeculae), cortical microarchitecture (total surface, polar moment of inertia), volumetric density of total, cortical and trabecular bone. Biological parameters: PTH, serum calcium and phosphorus, 25(OH)D, 1,25(OH)2D, biomarkers of bone remodelling, and urinary calcium. BMD measured by DXA. Clinical factor risks of bone loss.

Type of study : Pathophysiological, multicentric, comparative study, with a prospective follow-up of one year in postmenopausal caucasian women affected with PHPT (cases) or non affected by PHPT (controls). Each control will be matched for age, date of menopause, height and weight, to PHPT women.

Study design: assessment of bone and mineral metabolism, DXA and measurement of indices by HR-pQCT at the inclusion. Those tests will be renewed one year after surgery for the PHPT patients and one year after baseline for those without surgery and the controls.

Number of patients needed: 120 postmenopausal women, 60 cases and 60 controls

Total duration of the study: 56 months. Inclusion period : 42 months

Inclusion criteria and principal non-inclusion criteria :

Patients: caucasian women, menopaused for at least one year, aged less than 81 years, affected with symptomatic or asymptomatic PHPT and without any other disease or medication interfering with bone and mineral metabolism. Control population: caucasian women, menopaused for at least one year, aged less than 81 years, without PHPT, diseases or medications interfering with bone and mineral metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients: caucasian women, menopaused for at least one year, aged less than 81 years, affected with symptomatic or asymptomatic PHPT
* Control population: caucasian women, menopaused for at least one year, aged less than 81 years, without PHPT

Exclusion Criteria:

* diseases or medications interfering with bone and mineral metabolism

Max Age: 81 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cortical thickness measured by HR-pQCT | one year

SECONDARY OUTCOMES:
Three-dimensional evaluation of the cortical and trabecular bone by HR-pQCT | one year
Biological and quantitative parameters (assessed by HR-pQCT) | one year
Clinical, biological and bone densitometry parameters (assessed by DXA) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gerard MARUANI, MD, Principal Investigator — Hopital Europeen Georges Pompidou (HEGP)
Locations (3):
- France (3):
  - Hopital Lariboisiere, Paris
  - Hopital Cochin, Paris
  - Hopital Europeen Georges Pompidou, Paris